CLINICAL TRIAL: NCT04115566
Title: Hidradenitis Suppurativa Prospective Observational Registry and Biospecimen Repository
Acronym: HS PROGRESS
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 18-27002
Record Dates: First submitted 2019-09-18; First posted 2019-10-04 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hidradenitis suppurativa (HS) is a common and debilitating skin disease that is poorly understood and understudied. As a result, little is known about disease prognosis and few effective treatments exist for this condition. This prospective observational cohort study aims to comprehensively characterize the clinical and biological features of HS. The results of this research will provide a basis for the development of an HS clinical classification system and identification of potential treatments for HS.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 10 years of age
2. Diagnosis of HS by a dermatologist or practitioner experienced in making a diagnosis of HS
3. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Inability to give informed consent or unavailability of a parent/guardian who is able and willing to give informed consent.

Min Age: 10 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: HS Patients
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 2019-2029
  The primary aim of this study is to identify clinical and biologic characteristics of hidradenitis suppurativa.

SECONDARY OUTCOMES:
Secondary Objective | 2019-2029
  Secondary aims include correlating alterations in clinical and biological characteristics with disease status, and identifying genetic variants that predict disease progression or response to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Haley B Naik, MD, MHSc, FAAD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No